CLINICAL TRIAL: NCT00087386
Title: Phase II Trial of 17-N-allylamino-17-demethoxy Geldanamycin (17-AAG, NSC #330507) Diluted in EPL Diluent (NSC #704057) in Metastatic Melanoma Patients
Brief Title: Tanespimycin in Treating Patients With Stage III-IV Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01453; 04-056; NCI-6480; CDR0000374980; MSKCC-04056; N01CM62206 (NIH)
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Recurrent Melanoma; Stage III Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — tanespimycin

ARMS (1):
- Treatment (tanespimycin) (Experimental): Patients receive tanespimycin IV over 1-6 hours once weekly for 6 weeks. Courses repeat every 56 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tanespimycin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: tanespimycin — Given IV
  Other Names: 17-AAG
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well tanespimycin works in treating patients with stage III or stage IV melanoma. Antitumor antibiotics such as tanespimycin may stop the growth of melanoma by stopping blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine if treatment with 17-AAG results in measurable anti-tumor effects and calculate the proportion of clinical responses.

II. Test the hypothesis that treatment with 17-AAG can disrupt the MAPK pathway by depleting intra-tumor stores of RAF kinases and/or downstream proteins such as phospho-ERK, CDK4 and cyclin D1.

III. Determine if either of these effects correlates with the presence of mutated BRAF within the melanoma tumor.

OUTLINE: This is a multicenter study. Patients are stratified according to presence of BRAF mutation in tumor (yes vs no).

Patients receive tanespimycin IV over 1-6 hours once weekly for 6 weeks. Courses repeat every 56 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed melanoma

  * Stage III or IV disease
* No primary melanoma of the choroid or mucosa
* Measurable disease

  * At least 1 unidimensionally measurable lesion >= 20 mm by conventional techniques OR >= 10 mm by spiral CT scan
* Tumor amenable to biopsy (for the first 10 patients in each stratum only)

  * Patients must have measurable disease in addition to the tumor(s) to be biopsied
* No brain or epidural metastases

  * Completely resected solitary brain metastases allowed provided patient has been free of CNS metastases for >= 6 months
* Performance status - Karnofsky 60-100%
* Performance status - ECOG 0-2
* More than 3 months
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* WBC >= 3,000/mm^3
* AST and ALT =< 2.5 times upper limit of normal
* Creatinine normal
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No history of myocardial infarction
* No history of prolonged QTc interval
* No active ischemic heart disease within the past 12 months
* No uncontrolled dysrhythmia or dysrhythmias requiring medication
* No congenital prolonged QT syndrome
* No left bundle branch block
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to 17-N-allylamino-17-demethoxygeldanamycin (17-AAG)
* No prior serious allergic reaction to eggs
* No other uncontrolled illness
* No active or ongoing infection requiring systemic antimicrobial treatment
* No psychiatric illness or social situation that would preclude study compliance
* No more than 1 prior chemotherapy regimen for metastatic melanoma

  * Prior vaccines, cytokines, or interferon alfa is not considered prior therapy unless administered with a chemotherapy drug
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* Prior radiotherapy dose =< 3,000 cGy to fields including substantial marrow
* More than 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy field that included the heart (e.g., mantle)
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent medications that may prolong the QTc interval
* No other concurrent anticancer therapy
* No other concurrent investigational agents
* No concurrent treatment with any of the following medications or herbal remedies:

  * Inhibitors of CYP3A4:

    * Fluconazole
    * Itraconazole
    * Ketoconazole
    * Macrolide antibiotics (azithromycin, clarithromycin, erythromycin, or troleandomycin)
    * Midazolam
    * Nifedipine
    * Verapamil
    * Diltiazem
    * Terfenadine
    * Cyclosporine
    * Cisapride
  * Inducers of CYP3A4:

    * Carbamazepine
    * Phenobarbital
    * Phenytoin
    * Rifampin
  * Herbal extracts and tinctures with CYP3A4 inhibitory activity:

    * Hydrastis canadensis (goldenseal)
    * Hypericum perforatum (St. John's wort)
    * Uncaria tomentosa (cat's claw)
    * Echinacea angustifolia roots
    * Trifolium pratense (wild cherry)
    * Matricaria chamomilla (chamomile)
    * Glycyrrhiza glabra (licorice)
    * Dillapiol
    * Hypericin
    * Naringin
* No other concurrent herbal extracts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-06; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Response rate (complete and partial response) | Up to 3 years

SECONDARY OUTCOMES:
Proportion of patients with stable disease | At 1 year
Frequency of toxicities | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chapman, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States